CLINICAL TRIAL: NCT06073535
Title: The Usefulness of Injectable-Platelet Rich Fibrin in the Lower Third Molar Extraction: a Randomized-controlled Clinical Study.
Brief Title: The Use of Injectable-Platelet Rich Fibrin (i-PRF) in the Lower Third Molar Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Gilberto Sammartino, Full Professor, University of Naples
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UNaples
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Molar, Third; Postoperative Complications
Keywords: Molar, third; Postoperative complications; Swelling; Pain; Platelet-rich fibrin
MeSH Terms: conditions — Postoperative Complications; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator will be unaware of their treatment allocation before surgery. One clinician, not involved in patient treatment and not aware of what therapeutic approach, performed clinical measurement of face swelling on the surgery, 3th and 7th days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-PRF (Experimental): i-PRF will be used after the extraction of the third molar to reduce postoperative complications (swelling, pain) and wound healing.
  Interventions: Procedure: Extraction of mandibular third molar; Device: i-PRF
- Spontaneous healing (Active Comparator): After the extraction of the lower third molar the socket will be left to heal spontaneously.
  Interventions: Procedure: Extraction of mandibular third molar

INTERVENTIONS:
Procedure: Extraction of mandibular third molar — After loco-regional anesthesia was administered, a full-thickness mucoperiosteal flap was raised. The flap incision was extended from the vestibular side of the retromolar trigon to the second molar, corresponding to its distolingual cusp. The incision continued intrasulcular at the second molar and proceeded with a release incision distally to the papilla between the first and second molars, on a 45° angle.
  An osteotomy using a Lindemann burr under constant irrigation, followed by an odontotomy using a diamond burr was performed, if necessary.
Device: i-PRF — 20 ml of venous blood will be drawn from the ante-cubital vein of all patients and collected in 2 plastic tubes (Vacutainer, Becton& Dickinson, Rutherford, NJ) containing no anticoagulant or gelling agent. The tubes will be placed in a centrifuge (DUO Centrifuge, Nice, France) at 700 round per minute for 3 min, at the end of which time the blood will be separated into 2 fractions: the layer of injectable liquid i-PRF, which is more superficial, and the layer of red blood cells, in the deep part. From each tube, i-PRF will be withdrawn using a sterile syringe and it will be infiltrated into the lesion.
  Arms: i-PRF

SUMMARY:
Lower third molar extraction is one of the most frequently performed surgical procedures in dentistry. Common sequelae, including pain, swelling and trismus, can severely affect patients' quality of life during the immediate postoperative period.

The aim of this randomized-controlled trial is to clinically evaluate the reduction of lower third molar extraction-related complications, such as swelling and pain, and wound healing, following submucosal infiltration of injectable platelet rich fibrin.

DETAILED DESCRIPTION:
Forty young patients with a partially or totally impacted lower third molar, with an equivalent degree of difficulty, will be selected. All patients will be randomly treated by using 2 different therapeutic approaches, thereby yielding 2 different study groups, each of which is composed of 20 cases: in the first group, the extraction socket will be left healing spontaneously, while in the other side the socket will be filled with i-PRF.

This study was designed as a double-blind research since the investigator will be unaware of their treatment allocation before surgery, and one clinician, not involved in patient treatment and not aware of what therapeutic approach used for the different sites of treatment, will perform clinical measurement of the outcomes on the surgery day, 3th and 7th days after surgery.

A software will be used to produce a random sequence of 20 integer numbers without duplicates generated from atmospheric noise and concealed in closed envelopes by one of the investigators. At the time of the patient's first surgery, the envelope will be opened and patient allocated to group 1 or group 2.

Prior to surgery, photographic documentation consisting of frontal extraoral photograph, extraoral latero-lateral photograph of the surgery site, extraoral latero-lateral photograph of the opposite site will be performed.

The swelling will be measured summing two linear measurements of distance between Tragus and Pogonion and then Gonion and Commissura labialis points.

Immediately after surgery, the surgeon opens the envelope containing the information about the patient's group membership. In case of i-PRF group, 20 mL will be prepared.

Everyday after surgery, each patients will compile the visual analogic scale to evaluate the pain score.

On 3th and 7th day after surgery, linear measurements of swelling will be taken. Then, on 3th, 7th, 14th, 28th days the wound healing index by Landry will be evaluate.

The Student t test will be used to compare the differences between the two analysed groups. Potential differences between pain, swelling and wound healing based on gender, age and time of surgery will be assessed by using Student's t-test and one-way analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Need for extraction of totally or partially impacted lower third molar
* Equivalent degree of difficulty of lower third molar extraction
* Patients able to understand and sign informed consent

Exclusion Criteria:

* General contra-indications for surgery (systemic disease, compromised immune system etc);
* Tobacco smoking
* Alcohol and drug abuse
* Pregnancy and breastfeeding
* Patients taking any medications which might interfere with healing
* Dysplastic processes in the affected tooth elements
* Non-cooperative patients

EXCLUSION CRITERIA DURING FOLLOW-UP - Patients who do not adhere throughout the duration of follow-up to the specialist visits

POSTOPERATIVE EXCLUSION CRITERIA

- Taking more than two doses of prescribed anti-inflammatory/analgesic medication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Postoperative swelling | Measurements will be taken before surgery, on day 3 and day 7.
  Measurements will be made with a flexible ruler taking as reference the diagonals joining Tragus and Pogonion; Gonion and Labial Commissura. Swelling will be calculated as the sum of these diagonals.

SECONDARY OUTCOMES:
Postoperative pain | Everyday after surgery until 7th day.
  Pain was assessed with a visual analogic scale (VAS) from 0 (absence of pain) to 10 (severe pain).

OTHER OUTCOMES:
Wound healing | Measurements will be taken on day 3, 7, 14, 28 days.
  Landry index including description from a "Very poor" to an "Excellent" wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Sammartino, Professor, Principal Investigator — Federico II University
Locations (1):
- Gilberto Sammartino, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sammartino G, Gasparro R, Marenzi G, Trosino O, Mariniello M, Riccitiello F. Extraction of mandibular third molars: proposal of a new scale of difficulty. Br J Oral Maxillofac Surg. 2017 Nov;55(9):952-957. doi: 10.1016/j.bjoms.2017.09.012. Epub 2017 Oct 18. PMID 29054564
- [Result] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Result] Passaretti F, Tia M, D'Esposito V, De Pascale M, Del Corso M, Sepulveres R, Liguoro D, Valentino R, Beguinot F, Formisano P, Sammartino G. Growth-promoting action and growth factor release by different platelet derivatives. Platelets. 2014;25(4):252-6. doi: 10.3109/09537104.2013.809060. Epub 2013 Jul 15. PMID 23855408
- [Result] Dohan Ehrenfest DM, Bielecki T, Del Corso M, Inchingolo F, Sammartino G. Shedding light in the controversial terminology for platelet-rich products: platelet-rich plasma (PRP), platelet-rich fibrin (PRF), platelet-leukocyte gel (PLG), preparation rich in growth factors (PRGF), classification and commercialism. J Biomed Mater Res A. 2010 Dec 15;95(4):1280-2. doi: 10.1002/jbm.a.32894. Epub 2010 Oct 5. No abstract available. PMID 20925082
- [Result] Farshidfar N, Jafarpour D, Firoozi P, Sahmeddini S, Hamedani S, de Souza RF, Tayebi L. The application of injectable platelet-rich fibrin in regenerative dentistry: A systematic scoping review of In vitro and In vivo studies. Jpn Dent Sci Rev. 2022 Nov;58:89-123. doi: 10.1016/j.jdsr.2022.02.003. Epub 2022 Mar 29. PMID 35368368